CLINICAL TRIAL: NCT04246138
Title: RCT Comparing Functional Outcomes for Navigated Kinematically Aligned TKR Versus Navigated Mechanically Aligned TKR
Brief Title: A Randomised Control Trial Comparing Functional Outcomes for Navigated Kinematically Aligned TKR Versus Navigated Mechanically Aligned TKR
Acronym: MaKKRO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hull University Teaching Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: IRAS project no is 234077
Record Dates: First submitted 2020-01-27; First posted 2020-01-29 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2024-10

CONDITIONS: Kinematical Alignment,Mechanical Alignment, Navigation

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: randomisation done by software
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- kinematically alignment (Active Comparator)
  Interventions: Procedure: alignment types
- mechanical alignment (Active Comparator)
  Interventions: Procedure: alignment types

INTERVENTIONS:
Procedure: alignment types — types of alignment mechanical versus kinematic of TKA to be studied

SUMMARY:
The overall aim of the study is to compare navigated kinematically aligned total knee replacements (KA TKR) with navigated mechanically aligned TKR (MA TKR) in terms of function and ROM

The objectives are therefore:

1. To compare the functional outcomes of KA TKR versus MA TKR performed using navigation technique
2. To compare ROM and alignment of knee in the two groups

DETAILED DESCRIPTION:
STUDY DESIGN

1. .subject recruitment Patients will be recruited from the outpatient clinic of some of the orthopaedic surgeons working at Hull and East Yorkshire NHS trust hospitals over 18-24 months period. The patients coming to new clinic during this period will be explained about the trial and explained about the two methods of TKR- kinematically aligned and mechanically aligned. The participants involved in this study will NOT be paid any remuneration. The procedure involved and the follow up details will be explained to the patient and patient information leaflets handed over to them. The consent will be obtained in the clinic, in the presence of a nurse and / or family members of the patient. In case of non-English speaking patients, an interpreter will be called to do the translation of the communication between doctor and the patient. The interpreter in such scenarios will have to sign on the consent form in addition to the patients. Patients will be given sufficient time to arrive at a decision. In case they want to think over this study, they will be given one month, after which a telephonic conversation will be conducted to reach a decision. Patients can sign the consent form in the clinic or on the day of the surgery. On the day of surgery, reconfirmation of the consent to participate in the trial will be undertaken. Patient will be free to come out of trial at any stage of the trial if they wish to do so. Patients with special needs (mentally ill, children, those suffering from dementia) will be excluded from the study.
2. .Source of patients Patients visiting orthopaedic elective clinic of 2-3 consultants will be selected for this study. The study will be carried out at Hull Royal Infirmary and Castle Hill Hospitals. Expected number of patients eligible for the trial is 130 (65 in each group of kinematically aligned knee and mechanically aligned knee). We expect that at least 95% patients will agree to the trial. One surgeon will perform all kinematically aligned TKR and other surgeons will perform all mechanically aligned TKR which will ensure that there is no change of clinical practice for any surgeons in terms of kinematic or mechanical alignment of the TKR .

5….Randomisation Patients will be randomised using research randomiser computer software (randomisation.com).{16}.This program is a pseudo random number generator. The numbers are generated by complex algorithm (seeded by computer clock) that gives the appearance of randomness. This will help us randomly assign our study population into the two groups. It is a single blinded study and patients will be blinded. Envelopes will be opened after clinic appointment and patients will be booked for surgery based on which group they get randomised to.

6….withdrawal of subjects Patients may be withdrawn at any stage of the follow up/trial. If any patient develops dementia, deep infection, fracture, failure of extensor mechanism or any other injury which affects their mobility or ability to make decision will be withdrawn from the study. Under such circumstances randomization codes may have to be broken. Also if the patients want to sought second opinion or continue the treatment outside the trust, the codes may have to be broken. The codes will be available with the inpatient secretaries and may be obtained from them after taking due permission from the investigators. There won't be a need to replace a subject in this matter. Only randomization might have to be adjusted accordingly. The withdrawn subjects will be followed up in the clinics of respective surgeons, till a suitable period when they can be discharged to the care of the GPs, unless and until the subjects wishes not to do so.

7…Study treatments

Mechanical alignment considers only the two-dimensional (2D) alignment of the limb and knee in the coronal or frontal plane. Followers of mechanically aligned TKR strive to cut the distal femur perpendicular to a line drawn from the centre of the femoral head to the centre of the knee - the mechanical axis of the femur - and cut the proximal tibia perpendicular to a line drawn from the centre of the knee to the centre of the ankle - the mechanical axis of the tibia. Most surgeons using navigational rechnique for mechanically aligned TKR will aim to perform proximal tibial and distal femoral bony resection at 90 degrees to the mechanical axis of the femur and tibia..

In navigated kinematically-aligned TKA, the surgeon strives to position the femoral and tibial components to resurface the knee and restore the natural joint lines in the arthritic knee. The goal of kinematically aligned TKA is to restore the natural difference in symmetry and varus/valgus laxity between 0° of extension and 90° of flexion of the normal knee. Proximal tibial resection is performed to achieve equal thickness of medial and lateral bony resection accounting for wear and thickness of the saw blade. This usually results in varus tibial resection. To prevent excessive varus , a maximum upper limit of tibial resection is set at 3-4 degrees. Posterior slope is measured on xrays. Using navigation data exactly same amount of posterior slope is recreated accounting for 3 degrees of slope already present in tibial poly liner with Columbus TKR system.

After recording femoral data on navigation system and gap measurements, femoral resection is planned to achieve equal medial and lateral gaps in full extension but slightly wider gap on lateral side in flexion.

Both groups will undergo patella resurfacing irrespective of condition of the patella to remove potential bias if the patellar resurfacing is performed only in selective cases.

8…General information Name of treatment….Total knee replacement Device…. Columbus TKR manufactured by Bbraun Licence information in the UK….. This implant is widely available in UK and has gone through necessary approvals and is licensed for use in UK. This implant has been used by both surgeons as part of their usual orthopaedic practice Intended benefits. Pain and improved function Potential risks……infection, bleeding, scars, stiffness, persisting pain/deformity, loosening , fractures, dislocations, DVT , myocardial infarctions, cement reactions, stroke , death, damage to blood vessels and /or nerves, anaesthesia related complications , damage to extensor mechanism.

9….use of treatment within the trial Mechanically aligned and kinematically aligned knee replacement has been used in patients with symptomatic osteoarthritis who have not benefitted from non arthroplasty options. The efficacy has been validated in various studies. It is an invasive procedure carried out in operation theatres under anaesthesia. . The radiation involved in this study will be in form of X-rays which will be taken immediately preoperative (full leg alignment view), post-operative (standard ap/lat view) and at 1 year follow up (full leg alignment view). After the completion of trial the patients will be followed up in the clinic of operative surgeon until a period where they can be discharged to the care of respective GPs.

10…subject and compliance of study treatment The compliance will be assessed by the visits at follow up. If there is any missed follow up appointment, postal reminder will be sent. If the patient does not attend follow up visit on the consecutive appointment, it will be considered as lost to follow ups and discharged from the clinic.

COMPLIANCE WILL BE MONITORED WITH the help of Lorenzo software, to know if they were lost for follow ups. At such times, we will record the reason for a missed follow up after they have been missed for follow ups.

Patients lost to follow ups will be withdrawn from the study and will be followed as routine follow ups in the clinic of operating surgeon, unless they wish to do so.

11…….medications List of medications permitted during the trial

* Analgesia
* Antibiotics
* dalteparin List of medications not permitted during the trial
* none 12…. efficacy assessments( study procedures to measure efficacy) The primary outcome measure is KOOS at 12months Secondary outcomes

  * Knee ROM and stability (pre-op and at 1 year postop)
  * Oxford knee society score
  * SF-12
  * EQ5D
  * VAS pain score
  * Time taken for operation (tourniquest time)
  * Pre and post op distal femoral ,proximal tibial slopes on xray
  * Pre and post-Operative limb alignment
  * Hip knee ankle angle
  * KOOS ( Waterson et al study)

    13…safety assessments (study procedures to measure efficacy) The surgical interventions performed in this trial are part and parcel of the routine practice of the surgeons. The safety parameters are same as standard knee replacement performed in the unit. If there are any unusual complications (not listed above in para……) or higher rate of any complications, it will be reported.

    14….safety reporting

The collection and reporting of data on adverse events and serious adverse events will be in accordance with ICH GCP and the Research Governance Framework 2005.

15….samples No tissue or fluid samples will be taken during this trial 16…Data collection

* Source of the data

  o patient questionnaires (new society knee score

  o patient notes,

  o electronic data( patient clinic letters)

  o procedure ( as recorded on Lorenzo)

  o radiographs
* Time point for collection o Before surgery( baseline score)

  o 6 weeks post op

  o 6months post op

  o 1year follow up
* Who will collect the data? Independent researcher/practice nurse/physiotherapist/trainees/specialist registrar/trust registrars will collect the data
* List any data collected which will be considered to be source data i.e. data that will be used
* Clinic letters
* How the data will be made anonymous use of patient's initials and study number only).
* Why the data are being collected Initial baseline data and follow up quantitative and qualitative data for analysis and comparison between the two study groups.
* Whether the data are gathered using a standardised tool (e.g. McGill pain score), by means of a procedure (in which case full details should be supplied). If a nonstandard tool is to be used, detail on reliability and validity should be given.

No tools will be used for data collection; goniometers (mechanical/digital/app based) will be used to check ROM

* What form the data will take Binary data will be selected. Hard copies of clinical scores / ROM
* Describe methods used to maximise completeness of data Patient will be contacted if they are lost to follow up and in the database such patients will be red dotted 18….source data

As a minimum, the following information will be recorded in patient's case notes for study visits or telephone contacts:

19….protocol deviations /serious breaches All deviations from the protocol or GCP will be recorded by investigators on Protocol Deviation Form for the trial available from R&D. A serious breach is likely to affect to a significant degree either the safety or physical or mental integrity of a trial subject or the scientific value of the trial. Major deviations or serious breaches will be reported by investigators to HEY R&D by telephone (tel 461883) or in person within 24 hours of the deviation or breach being identified. HEY R&D will notify the REC within 7 days of becoming aware of a serious breach. Investigators will take into account all protocol deviations and any serious breaches in the final study analysis and publication.

20….study equipment All the equipment's and implants used in the study are a part of routine knee replacement practice of both surgeons. The details of the implant. Confirmation that the implant will be available during the course of the study. The arrangements made for availability of the equipment, proper and timely maintenance and calibration of equipment.

21….end of trial The trial will end when the last patient participating in the trial will complete 1 year follow up.

In case of discontinuation of trial, an interim analysis will take place with the help of clinical director for orthopaedics.

An end of study declaration form (using the NRES form) will be submitted to the REC and Trust R&D within 90 days from completion of the trial and within 15 days if the trial is discontinued prematurely. A summary of the trial report/publication will be submitted to the REC and Trust R&D within 1 year of the end of trial 22….sample size calculation Waterson et al (17) found that at 12 months the mean KOOS score was 77.7 (20.0 sd) in the KA TKR group. This study is powered to demonstrate a 19 point difference in the KOOS score between groups at 12 months which has been defined as the minimal clinical important (MCI) difference in scores by the research team. Further literature review (20) confirms that the MCI for KOOS after TKR actually ranges from 11 to 19 for various sub categories of KOOS. As our study involves TKR as the main intervention it was agreed with the statistician to use the above MCI figures which are more relevant to our study. Hence sample size was recalculated for detecting a difference of 11 points for KOOS between 2 groups to ensure that study is sufficiently powered. New sample size of 42 in each group is now agreed with statistician assuming same standard deviation od 20 points in KOOS, using a one tailed analysis and an alpha of 0.05 with a power of 0.80

23….statistical analysis This trial will be reported according to the CONSORT guidelines for clinical trials (Consolidated Standards Of Reporting Trials statement (http://www.consort-statement.org/)). Analyses will be conducted following the principles of intention-to-treat with patient's outcomes analysed according to their original, randomised group irrespective of deviations based on non-compliance.

Analyses will be undertaken in Stata v14 or later (to be confirmed in the final report). Significance tests will be two-sided at the 5% significance levels unless otherwise stated. The statistician will remain blind to allocation until after the trial is complete and the results have been finalised.

The number of patients screened, eligible and randomised will be reported. The flow of participants through the trial will be presented in a CONSORT diagram. Questionnaire response rates will be summarised from each time point by treatment group.

All participant baseline data will be summarised descriptively overall and by trial arm both as randomised and as analysed in the primary analysis. No formal statistical comparisons will be undertaken. Continuous measures will be reported as means and standard deviations while the categorical data will be reported as counts and percentages.

The primary analysis will compare the KOOS at 12 months among the patients randomly allocated to KA TKR and MA TKR. This result will be extracted from a covariance pattern model in which KOOS at each time point (Baseline, 6 weeks , 6 months and 12 months) will be nested within patients and the effect of treatment according to trial arm will be assessed. KOOS at baseline, trial arm, each time point of follow-up, each time point of follow-up by trial arm interaction, any stratification factors (fixed effects) and KOOS at each time point nested within patient (random effects) will be included in the model. This will allow efficient use of the data collected, and account for potential correlation of repeated measures and within patient correlation.(18)

Different covariance structures for the repeated measurements, that are available as part of Stata, will be explored and the most appropriate pattern will be used for the final model. Diagnostics including Akaike's information criterion [19] will be compared for each model (smaller values are preferred).

Participants are included in the model if they have full data for the baseline covariates and outcome data for at least one post-randomisation time point. A comparison of baseline data for patients 'as analysed' in the primary analysis will allow assessment of whether attrition has introduced selection bias.

This linear mixed model will also provide an estimate of the comparable effect of KA TKR and MA TKR in terms of a change in KOOS at every time point for secondary investigations aimed at determining any potential pattern of improvement. Treatment effect sizes will be reported with 95% confidence intervals for each time point. The assumptions of the linear model will be checked visually. The normality of the standardised residuals will be assessed via a histogram and QQ-plot, and the homoscedasticity of the errors will be checked by plotting the residuals against the fitted valvalues. If model assumptions are in doubt, transformations will be considered.

Secondary outcome data will be summarised descriptively at each time point, overall and by trial arm and will be analysed in exactly the same way as the primary outcome.

24…pharmacy There is no role of pharmacy in the trial. The implants have been in use all over the UK and in the trust for more than 5 years and will be available for future use in the trust during the trial 25….Quality control and quality assurance

a…Peer review This trial has been Peer reviewed and discussed in clinical governance meeting of orthopaedic department by Name Mr T Symes Position clinical director, Orthopaedic department Address Hull Royal Infirmary, Anlaby Road, Hull, HU3 2JZ Contact details tom.symes@hey.nhs.uk b….monitoring The study may be monitored in accordance with HEY R&D department standard operating procedures to ensure compliance with ICH GCP and the Research governance Framework 2005. All trial related documents will be made available upon request for monitoring by R&D monitors

26….Ethical considerations The treatment modalities offered in the trial, are part and parcel of the surgeons routine knee replacement practice. Hence there are not obvious ethical considerations in this trial

ELIGIBILITY:
Inclusion Criteria:

* • Age between 18 and 90 years

  * Diagnosis of degenerative osteoarthritis

Exclusion Criteria:

* o a)Post traumatic arthritis

  * b)Varus /valgus deformity of more than 20 degrees

    * flexion contracture of more than 20 degrees
    * reduced ability to make decision like dementia patients/children
  * e)if they had undergone any orthopaedic procedure to the lower limbs within the last one year
  * h) neuromuscular or neurosensory deficiency
  * I)inflammatory arthritis of the knee joint

    * patients who suffered a complication which might influence the final outcome such as a deep infection, fracture or dysfunction of the extensor mechanism in post-operative period. However the complication rate data will be analysed and reported.
    * pregnancy
    * patients involved in other clinical trials within last 6 months prior to being recruited in the study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-02-18 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
KOOS | 12 months
  knee osteoarthritis outcome score preop and at 12 months

SECONDARY OUTCOMES:
• Knee ROM and stability (pre-op and at 1 year postop) | 1 year
  to be checked by independent assessor
• Oxford knee society score | 1 year
  patient based outcomes
• SF-12 | 1 year
  patiuent based outcomes
• EQ5D | 1 year
• Time taken for operation (tourniquest time) | 1 year
  from operation notes
Pre and post op DFA,tibial slope on xray • • Pre and post op distal femoral ,proximal tibial slopes on xray • • Pre and post op distal femoral ,proximal tibial slopes on xray • • Pre and post op distal femoral ,proximal tibial slopes on xray | 1 year
  measured on xray
• Pre and post-Operative limb alignment | 1 year
  measured on xray
• Hip knee ankle angle | 1 year
  on xray

CONTACTS AND LOCATIONS:
Locations (1):
- Hull University teaching hospitals, Hull, East Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No